CLINICAL TRIAL: NCT02387398
Title: A Pilot Randomized Clinical Trial of Early Coronary Angiography Versus No Early Coronary Angiography for Post-Cardiac Arrest Patients Without ECG ST Segment Elevation
Brief Title: Early Coronary Angiography Versus Delayed Coronary Angiography
Acronym: PEARL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funded study period, including a one-year no cost extension, completed.
Sponsor: University of Arizona (Other)
Collaborators: MaineHealth (Other); University Medical Centre Ljubljana (Other); Mayo Clinic (Other); The Alfred (Other)
Responsible Party: Principal Investigator, Karl Kern, MD, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT02387398
Record Dates: First submitted 2015-02-26; First posted 2015-03-13 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Out-of-Hospital Cardiac Arrest; Hypothermia; Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypothermia; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional (Experimental): Early Angiography with purpose of coronary revascularization within 120 minutes of admission to ED, post out-of-hospital cardiac arrest, suspicious for cardiac etiology and no ST segment elevation on ECG
  Interventions: Procedure: Early Angiography
- Control Group (No Intervention): Standard of care treatment including therapeutic hypothermia in subjects post resuscitation, out-of-hospital cardiac arrest, suspicious for cardiac etiology and no ST segment elevation on ECG.

INTERVENTIONS:
Procedure: Early Angiography — Coronary Angiography within 120 minutes of admission for out-of-hospital cardiac arrest with ROSC
  Arms: Interventional

SUMMARY:
This study is a pilot, multi-centered, randomized, clinical trial to evaluate the safety and efficacy of performing early Coronary Angiography (CAG) versus no early CAG in post-cardiac arrest patients without ST segment elevation. Safety will be assessed by evaluating the association of major adverse events (re-arrest, bleeding, pulmonary edema, hypotension, acute renal insufficiency, and pneumonia) with early coronary angiogram. Efficacy will be assessed by a composite endpoint of improved left ventricular regional and global function (both regional wall motion analysis and left ventricular ejection fraction) as measured by echocardiography prior to hospital discharge and favourable neurological function (Cerebral Performance Categories 1 or 2) at discharge.

DETAILED DESCRIPTION:
Cardiac arrest is a major public health issue. Arizona has been a leader in improving long-term survival by introducing new and innovative resuscitation approaches including "Chest Compression-Only CPR" and "Cardiocerebral Resuscitation". Post-resuscitation care is the next great opportunity for further improvements. Early coronary angiography (CAG) combined with therapeutic hypothermia has become the recommended standard of care for post-cardiac arrest patients manifesting ST segment elevation on their electrocardiogram (ECG). However, the majority of cardiac arrest victims do not have ST segment elevation. There is clinical equipoise as to whether these patients will benefit from early CAG.

Subjects who are qualified for the study will be randomized 1:1 to one of two groups.

° Intervention Group-Early coronary angiography (door-to-angiography) within 120 minutes of admission to Emergency Department.

or

° Control Group-No early coronary angiography (within the first six hours from admission)

All enrolled patients, will be treated with therapeutic hypothermia which is standard of care, beginning simultaneously with both groups or within at least 2 hours of hospital arrival.

Subject will be followed for 180 days for safety and long-term survival.

ELIGIBILITY:
Inclusion Criteria:

1. All successfully resuscitated out-of-hospital cardiac arrest patients with a suspected cardiac etiology for their non-traumatic arrest
2. Age greater than 18 years
3. The post resuscitation ECG shows no evidence of ST segment elevation

Exclusion Criteria:

1. Non-resuscitated (no sustained pulse and BP)
2. Presence ST segment elevation or new left bundle branch block present on the post-resuscitation ECG
3. Suspected non-cardiac etiology for their arrest such as respiratory failure, asphyxia, pulmonary embolus, shock, trauma, drug overdose, or CNS bleed as likely cause of the cardiac arrest
4. Known "Do Not Resuscitate" status
5. Minors (<18 years old)
6. Prisoners
7. Significant bleeding or blunt trauma
8. Known or confirmed pregnancy test by urinalysis
9. Patients who are known to have received any other investigational therapies within the 30 days prior to enrollment or during study duration will be excluded unless these studies have been reviewed and approved by the Study Steering Committee.
10. Known "opt out" choice; wearing Opt-out band for any EFIC approved study or on an "Opt-out" list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of early coronary angiography in the out-of-hospital cardiac arrest (OHCA) patient population. | 180 days
  Safety will be assessed by evaluating any association of major adverse events (re-arrest, bleeding, pulmonary edema, hypotension, acute renal insufficiency, and pneumonia) with early coronary angiography.

SECONDARY OUTCOMES:
Survival from hospital at: 30 days post discharge and 180 days post discharge | 30 days and 180 days
  Composite endpoint of improved left ventricular regional and global function (both regional wall motion analysis and left ventricular ejection fraction) as measured by echocardiography prior to hospital discharge, survival to discharge and favourable. Left ventricular regional function and left ventricular ejection fraction as measured by echocardiography will be measured prior to discharge or up to 180 days post hospital discharge.
Cognitive functional status | 180 days
  As measured by Modified Rankin Score (mRS) and Cerebral Performance Category (CPC) at multiple points up to 180 days post hospital discharge
Neurocognitive Testing | 180 days
  Neurocognitive function will be assessed at various time points utilizing a variety of tests from ICU discharge to 180 days post hospital discharge such as MMSE, MOCA, HADS, and IQCODE

CONTACTS AND LOCATIONS:
Overall Officials: Karl B Kern, MD, Principal Investigator — University of Arizona
Locations (6):
- United States (4):
  - Banner University Medical Center-South Campus, Tucson, Arizona
  - Banner University Medical Center-Tucson Campus, Tucson, Arizona
  - Tufts University School of Medicine, Maine Medical Center, Portland, Maine
  - Mayo Clinic Cardiovascular Research Unit, Rochester, Minnesota
- Alfred Hospital, Melbourne, Victoria, Australia
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kern KB, Radsel P, Jentzer JC, Seder DB, Lee KS, Lotun K, Janardhanan R, Stub D, Hsu CH, Noc M. Randomized Pilot Clinical Trial of Early Coronary Angiography Versus No Early Coronary Angiography After Cardiac Arrest Without ST-Segment Elevation: The PEARL Study. Circulation. 2020 Nov 24;142(21):2002-2012. doi: 10.1161/CIRCULATIONAHA.120.049569. Epub 2020 Sep 28. PMID 32985249